CLINICAL TRIAL: NCT03371628
Title: Use of Electrical Impedance Tomography in Evaluating the Effects of Noninvasive Ventilation in the Post-Operative Cardiac Surgery: Controlled and Randomized Clinical Trial
Brief Title: Electrical Impedance Tomography in Evaluating the Effects of Noninvasive Ventilation in Post-Operative Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Alita Paula Lopes de Novaes, Master´s program studant, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tomografia de Impedância
Record Dates: First submitted 2017-11-20; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Thoracic Surgery
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: A parallel group study is a simple and commonly used clinical design which compares two treatments. Usually a test therapy is compared with a standard therapy. The allocation of subjects to groups is usually achieved by randomisation. The groups are typically named the treatment group and the control group. Parallel group designs do not require the same number of subjects in each group, although often similar numbers are observed. The design is commonly used in randomised controlled trials. Statistical analysis often boils down to a simple t-test of the between group difference in the outcome, which is usually a mean or a proportion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group VNI 1h (Experimental): Intervention: Non invasive ventilation, applied for 1 hour
  Interventions: Device: Non invasive ventilation
- Group O2 (No Intervention): Oxygen therapy

INTERVENTIONS:
Device: Non invasive ventilation — Non invasive ventilation is a mode of mechanical ventilation that does not require the use of artificial airway.
  Arms: Group VNI 1h

SUMMARY:
NTRODUCTION: cardiac surgery can lead to pulmonary complications such as hypoxemia and atelectasis. Noninvasive ventilation has been used to prevent and treat such complications. Electrical impedance tomography has been a useful tool in bedside evaluation of ventilation and pulmonary ventilation. OBJECTIVE: To compare the effects of non-invasive ventilation with oxygen therapy in cardiac post-operative patients. MATERIALS AND METHODS: It will be a randomized controlled clinical trial where patients will be divided into two groups: a group that will perform NIV for 1 hour and the group that will only use oxygen therapy. They will be evaluated through Electrical Impedance Tomography and arterial gasometry analysis just before extubation, soon after extubation, during the intervention and after the intervention for a period of 2 hours after extubation. EXPECTED RESULTS: It is expected that the NIV group will present higher pulmonary ventilation and aeration and better gas exchange than the oxygen therapy group, and that the time of therapeutic effect will be higher in the NIV group.

DETAILED DESCRIPTION:
The proposal basically consists of Validation of the hypothesis: The use of Non-invasive Ventilation in patients in the postoperative cardiac surgery results in greater ventilation, greater aeration, and improved gas exchange when compared to the oxygen therapy group.

The use of noninvasive ventilation in the postoperative cardiac surgery has been widely used in clinical practice, but the evidence of the benefits of this technique in this population in relation to some criteria have not yet been elucidated in the scientific literature, such as the effect of NIV in ventilation and pulmonary ventilation, and how long does this effect last.

ELIGIBILITY:
Inclusion Criteria:

* Immediate postoperative period of cardiac surgery
* age between 18 and 65 years
* BMI between 18.5 and 30 kg / m2
* Patients still intubated when admitted to the ICU
* without previous history of severe pulmonary diseases such as chronic obstructive pulmonary disease, pulmonary fibrosis, or chronic renal failure, or associated neuromuscular diseases

Exclusion Criteria:

* Patients considered to be at risk for extubation failure (hypercapnia, more than failure in the autonomic test, AVM time greater than 72 hours, ineffective cough)
* Cardiopulmonary bypass time more than 150 minutes
* Hemodynamic instability (arrhythmias, cardiogenic shock, severe hypotension with SBP <90mmHg)
* Episodes of abdominal distension, nausea and vomiting
* Hypoxemia (PO2 <50mmHg with FiO2 50%) or hypercapnia (PaCO2> 55mmHg with pH <7.30)
* Patients who are at high surgical risk according to Euroscore II

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2017-12-06 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
change in electrical impedance measures | data recorded 5 minutes before extubation, 5 minutes after extubation, at the first 5 minutes of therapy, 25 to 30 minutes after beginning of therapy, 55 to 60 minutes after beginning of therapy, and 1,5 hour and 2 hours after beginning of therapy
  impedance variation data recorded by impedance electrical tomography

SECONDARY OUTCOMES:
change in Blood gases analysis - PaO2 (mmHg), PaCO2 (mmHg), PaO2/FiO2 | recorded 5 minutes before extubation and 1 hour after extubation
  Collected by a Laboratory professional

CONTACTS AND LOCATIONS:
Overall Officials: Daniella C Brandão, PhD, Study Director — UFPE
Locations (1):
- Alita Paula Lopes de Novaes, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Datas relative to the results of the use of electrical impedance tomography, besides blood gases and vital signs.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: march 2018
Access Criteria: Date will be available by a USB pen drive copy by the researchers, including date relative to electrical impedance tomography and to bloog gases

REFERENCES:
- [Background] Jaber S, Chanques G, Jung B. Postoperative noninvasive ventilation. Anesthesiology. 2010 Feb;112(2):453-61. doi: 10.1097/ALN.0b013e3181c5e5f2. No abstract available. PMID 20068454
- [Background] Rahmanian PB, Kroner A, Langebartels G, Ozel O, Wippermann J, Wahlers T. Impact of major non-cardiac complications on outcome following cardiac surgery procedures: logistic regression analysis in a very recent patient cohort. Interact Cardiovasc Thorac Surg. 2013 Aug;17(2):319-26; discussion 326-7. doi: 10.1093/icvts/ivt149. Epub 2013 May 10. PMID 23667066
- [Background] Zarbock A, Mueller E, Netzer S, Gabriel A, Feindt P, Kindgen-Milles D. Prophylactic nasal continuous positive airway pressure following cardiac surgery protects from postoperative pulmonary complications: a prospective, randomized, controlled trial in 500 patients. Chest. 2009 May;135(5):1252-1259. doi: 10.1378/chest.08-1602. Epub 2008 Nov 18. PMID 19017864
- [Background] Diodato M, Chedrawy EG. Coronary artery bypass graft surgery: the past, present, and future of myocardial revascularisation. Surg Res Pract. 2014;2014:726158. doi: 10.1155/2014/726158. Epub 2014 Jan 2. PMID 25374960
- [Background] Niclauss L. Techniques and standards in intraoperative graft verification by transit time flow measurement after coronary artery bypass graft surgery: a critical review. Eur J Cardiothorac Surg. 2017 Jan;51(1):26-33. doi: 10.1093/ejcts/ezw203. Epub 2016 Jun 13. PMID 27298393
- [Background] Yazdannik A, Bollbanabad HM, Mirmohammadsadeghi M, Khalifezade A. The effect of incentive spirometry on arterial blood gases after coronary artery bypass surgery (CABG). Iran J Nurs Midwifery Res. 2016 Jan-Feb;21(1):89-92. doi: 10.4103/1735-9066.174761. PMID 26985228
- [Background] Al Jaaly E, Fiorentino F, Reeves BC, Ind PW, Angelini GD, Kemp S, Shiner RJ. Effect of adding postoperative noninvasive ventilation to usual care to prevent pulmonary complications in patients undergoing coronary artery bypass grafting: a randomized controlled trial. J Thorac Cardiovasc Surg. 2013 Oct;146(4):912-8. doi: 10.1016/j.jtcvs.2013.03.014. Epub 2013 Apr 11. PMID 23582830
- [Background] Kotani T, Tanabe H, Yusa H, Saito S, Yamazaki K, Ozaki M. Electrical impedance tomography-guided prone positioning in a patient with acute cor pulmonale associated with severe acute respiratory distress syndrome. J Anesth. 2016 Feb;30(1):161-5. doi: 10.1007/s00540-015-2084-y. Epub 2015 Oct 7. PMID 26446805
- [Background] Vogt B, Pulletz S, Elke G, Zhao Z, Zabel P, Weiler N, Frerichs I. Spatial and temporal heterogeneity of regional lung ventilation determined by electrical impedance tomography during pulmonary function testing. J Appl Physiol (1985). 2012 Oct;113(7):1154-61. doi: 10.1152/japplphysiol.01630.2011. Epub 2012 Aug 16. PMID 22898553
- [Background] Parolari A, Poggio P, Myasoedova V, Songia P, Bonalumi G, Pilozzi A, Pacini D, Alamanni F, Tremoli E. Biomarkers in Coronary Artery Bypass Surgery: Ready for Prime Time and Outcome Prediction? Front Cardiovasc Med. 2016 Jan 5;2:39. doi: 10.3389/fcvm.2015.00039. eCollection 2015. PMID 26779491
- [Background] Mendes RG, de Souza CR, Machado MN, Correa PR, Di Thommazo-Luporini L, Arena R, Myers J, Pizzolato EB, Borghi-Silva A. Predicting reintubation, prolonged mechanical ventilation and death in post-coronary artery bypass graft surgery: a comparison between artificial neural networks and logistic regression models. Arch Med Sci. 2015 Aug 12;11(4):756-63. doi: 10.5114/aoms.2015.48145. Epub 2015 Aug 11. PMID 26322087
- [Background] Kochamba GS, Yun KL, Pfeffer TA, Sintek CF, Khonsari S. Pulmonary abnormalities after coronary arterial bypass grafting operation: cardiopulmonary bypass versus mechanical stabilization. Ann Thorac Surg. 2000 May;69(5):1466-70. doi: 10.1016/s0003-4975(00)01142-5. PMID 10881824
- [Background] Chiumello D, Chevallard G, Gregoretti C. Non-invasive ventilation in postoperative patients: a systematic review. Intensive Care Med. 2011 Jun;37(6):918-29. doi: 10.1007/s00134-011-2210-8. Epub 2011 Mar 18. PMID 21424246
- [Background] Glossop AJ, Shephard N, Bryden DC, Mills GH. Non-invasive ventilation for weaning, avoiding reintubation after extubation and in the postoperative period: a meta-analysis. Br J Anaesth. 2012 Sep;109(3):305-14. doi: 10.1093/bja/aes270. PMID 22879654
- [Background] Perrin C, Jullien V, Venissac N, Berthier F, Padovani B, Guillot F, Coussement A, Mouroux J. Prophylactic use of noninvasive ventilation in patients undergoing lung resectional surgery. Respir Med. 2007 Jul;101(7):1572-8. doi: 10.1016/j.rmed.2006.12.002. Epub 2007 Jan 25. PMID 17257820
- [Background] Olper L, Corbetta D, Cabrini L, Landoni G, Zangrillo A. Effects of non-invasive ventilation on reintubation rate: a systematic review and meta-analysis of randomised studies of patients undergoing cardiothoracic surgery. Crit Care Resusc. 2013 Sep;15(3):220-7. PMID 23944209
- [Background] Becher T, Vogt B, Kott M, Schadler D, Weiler N, Frerichs I. Functional Regions of Interest in Electrical Impedance Tomography: A Secondary Analysis of Two Clinical Studies. PLoS One. 2016 Mar 24;11(3):e0152267. doi: 10.1371/journal.pone.0152267. eCollection 2016. PMID 27010320
- [Background] Victorino JA, Borges JB, Okamoto VN, Matos GF, Tucci MR, Caramez MP, Tanaka H, Sipmann FS, Santos DC, Barbas CS, Carvalho CR, Amato MB. Imbalances in regional lung ventilation: a validation study on electrical impedance tomography. Am J Respir Crit Care Med. 2004 Apr 1;169(7):791-800. doi: 10.1164/rccm.200301-133OC. Epub 2003 Dec 23. PMID 14693669
- [Background] Frerichs I, Dargaville PA, Dudykevych T, Rimensberger PC. Electrical impedance tomography: a method for monitoring regional lung aeration and tidal volume distribution? Intensive Care Med. 2003 Dec;29(12):2312-2316. doi: 10.1007/s00134-003-2029-z. Epub 2003 Oct 18. PMID 14566457
- [Background] Costa EL, Chaves CN, Gomes S, Beraldo MA, Volpe MS, Tucci MR, Schettino IA, Bohm SH, Carvalho CR, Tanaka H, Lima RG, Amato MB. Real-time detection of pneumothorax using electrical impedance tomography. Crit Care Med. 2008 Apr;36(4):1230-8. doi: 10.1097/CCM.0b013e31816a0380. PMID 18379250
- [Background] Costa EL, Borges JB, Melo A, Suarez-Sipmann F, Toufen C Jr, Bohm SH, Amato MB. Bedside estimation of recruitable alveolar collapse and hyperdistension by electrical impedance tomography. Intensive Care Med. 2009 Jun;35(6):1132-7. doi: 10.1007/s00134-009-1447-y. Epub 2009 Mar 3. PMID 19255741
- [Background] Stankiewicz-Rudnicki M, Gaszynski T, Gaszynski W. Assessment of regional ventilation in acute respiratory distress syndrome by electrical impedance tomography. Anaesthesiol Intensive Ther. 2015;47(1):77-81. doi: 10.5603/AIT.2015.0007. PMID 25751294
- [Background] Leonhardt S, Lachmann B. Electrical impedance tomography: the holy grail of ventilation and perfusion monitoring? Intensive Care Med. 2012 Dec;38(12):1917-29. doi: 10.1007/s00134-012-2684-z. Epub 2012 Sep 20. PMID 22992946
- [Background] Karsten J, Grusnick C, Paarmann H, Heringlake M, Heinze H. Positive end-expiratory pressure titration at bedside using electrical impedance tomography in post-operative cardiac surgery patients. Acta Anaesthesiol Scand. 2015 Jul;59(6):723-32. doi: 10.1111/aas.12518. Epub 2015 Apr 13. PMID 25867049
- [Background] Blankman P, Shono A, Hermans BJ, Wesselius T, Hasan D, Gommers D. Detection of optimal PEEP for equal distribution of tidal volume by volumetric capnography and electrical impedance tomography during decreasing levels of PEEP in post cardiac-surgery patients. Br J Anaesth. 2016 Jun;116(6):862-9. doi: 10.1093/bja/aew116. PMID 27199318
- [Background] Tanaka H, Ortega NR, Galizia MS, Borges JB, Amato MB. Fuzzy modeling of electrical impedance tomography images of the lungs. Clinics (Sao Paulo). 2008 Jun;63(3):363-70. doi: 10.1590/s1807-59322008000300013. PMID 18568247
- [Background] Kobylianskii J, Murray A, Brace D, Goligher E, Fan E. Electrical impedance tomography in adult patients undergoing mechanical ventilation: A systematic review. J Crit Care. 2016 Oct;35:33-50. doi: 10.1016/j.jcrc.2016.04.028. Epub 2016 May 3. PMID 27481734
- [Background] Landoni G, Zangrillo A, Cabrini L. Noninvasive ventilation after cardiac and thoracic surgery in adult patients: a review. J Cardiothorac Vasc Anesth. 2012 Oct;26(5):917-22. doi: 10.1053/j.jvca.2011.06.003. Epub 2011 Aug 11. No abstract available. PMID 21835640
- [Background] Bordes J, Goutorbe P, Cungi PJ, Boghossian MC, Kaiser E. Noninvasive ventilation during spontaneous breathing anesthesia: an observational study using electrical impedance tomography. J Clin Anesth. 2016 Nov;34:420-6. doi: 10.1016/j.jclinane.2016.04.016. Epub 2016 Jun 16. PMID 27687426
- [Background] Zhai J, Wei L, Huang B, Wang C, Zhang H, Yin K. Minimally invasive mitral valve replacement is a safe and effective surgery for patients with rheumatic valve disease: A retrospective study. Medicine (Baltimore). 2017 Jun;96(24):e7193. doi: 10.1097/MD.0000000000007193. PMID 28614262
- [Background] Eronia N, Mauri T, Maffezzini E, Gatti S, Bronco A, Alban L, Binda F, Sasso T, Marenghi C, Grasselli G, Foti G, Pesenti A, Bellani G. Bedside selection of positive end-expiratory pressure by electrical impedance tomography in hypoxemic patients: a feasibility study. Ann Intensive Care. 2017 Dec;7(1):76. doi: 10.1186/s13613-017-0299-9. Epub 2017 Jul 20. PMID 28730554
- [Background] Yildirim F, Esquinas AM, Glossop AJ. Noninvasive mechanical ventilation during spontaneous breathing anaesthesia: Can electrical impedance tomography be a useful bedside tool to titrate PEEP level? J Clin Anesth. 2017 Jun;39:106-107. doi: 10.1016/j.jclinane.2017.03.030. Epub 2017 Apr 4. No abstract available. PMID 28494880